CLINICAL TRIAL: NCT05484271
Title: Relationship Between the Arthroscopic Anatomy of the Middle Glenohumeral Ligament and the Rotator Cuff Tear Position
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IIT-2022-0074
Record Dates: First submitted 2022-08-01; First posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Rotator Cuff Tears
Keywords: Rotator Cuff Tears; Middle Glenohumeral Ligament; Arthroscopic Anatomy
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Leaf-like and Cord-like type: Under arthroscopy, the anatomy of middle glenohumeral ligament was leaf-like or cord-like.
  Interventions: Procedure: Rotator cuff repair
- Absent type: Under arthroscopy, the anatomy of middle glenohumeral ligament was absent.
  Interventions: Procedure: Rotator cuff repair
- Burford complex type: Under arthroscopy, the anatomy of middle glenohumeral ligament manifested the burford complex.
  Interventions: Procedure: Rotator cuff repair

INTERVENTIONS:
Procedure: Rotator cuff repair — The patients received the arthroscopic rotator cuff repair.

SUMMARY:
The main aim and scope of this study is making observation and comparing the difference in the tear position in the patients suffered form rotator cuff tear with different arthroscopic anatomy of the middle glenohumeral ligament. The results may identify the influence of the middle glenohumeral ligament anatomy type on the rotator cuff tear.

ELIGIBILITY:
Inclusion Criteria:

* partial or full-thickness but reparable rotator cuff tear;
* small- to large-sized rotator cuff tears being defined by DeOrio and Cofied4;
* no improvements after at least 1 month of conservative treatment such as NSAIDs or corticosteroid injection.

Exclusion Criteria:

* massive rotator cuff tears being defined by DeOrio and Cofied;
* patients with osteoarthritis of the glenohumeral joint;
* trauma or a history of surgery at the shoulder.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with rotator cuff tears received the arthroscopic rotator cuff repair.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2022-08-05 (Estimated); Primary Completion 2022-08-20 (Estimated); Study Completion 2022-08-28 (Estimated)

PRIMARY OUTCOMES:
The arthroscopic tear position (Anetrior/Middle/Posterior) | During the surgery
  The rotator cuff was divided into three parts according to the arthroscopic discovery: (1) the anterior part which contained the subsacpularis and one third of the suprascapularis forward; (2) the middle part which contained the two thirds of the suprascapularis backward and one third of the subscapularis forward; (3) the posterior part which contained two thirds of subscapularis backward and teres minor.